CLINICAL TRIAL: NCT02159001
Title: Efficacy and Cognitive Effects of Electroconvulsive Therapy in Clozapine-Resistant Schizophrenia
Brief Title: Electroconvulsive Therapy in Clozapine-resistant Schizophrenia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Niuvanniemi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 22014
Record Dates: First submitted 2014-06-04; First posted 2014-06-09 (Estimated); Last update posted 2015-10-16 (Estimated); Status verified 2015-10

CONDITIONS: Schizophrenia; Schizoaffective Disorder
Keywords: clozapine; ECT; PANSS; schizoaffective disorder; schizophrenia; treatment
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ECT treatment right after recruitment (Active Comparator): This group receives electroconvulsive therapy treatment right after they are recruited.
  Interventions: Device: electroconvulsive therapy
- ECT after 4 weeks period. (Placebo Comparator): This group receives electroconvulsive therapy treatment after 4 weeks waiting period.
  Interventions: Device: electroconvulsive therapy

INTERVENTIONS:
Device: electroconvulsive therapy — 10-course, three times a week bilateral frontotemporal ECT

SUMMARY:
Electroconvulsive therapy (ECT) is one of the oldest neuromodulation treatments still used in psychiatry. Only case reports and open label non-randomized studies have been published of ECT in clozapine-resistant schizophrenia patients. The purpose of this trial is to study the efficacy and cognitive effects of add-on ECT treatment (10-course) in schizophrenia patients taking clozapine.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of schizophrenia or schizoaffective disorder
* treatment-resistant to clozapine
* age 18 - 64 years
* capacity and willingness to give informed consent

Exclusion Criteria:

* serious somatic illness
* progressive neurological illness, recent brain damage or sequela of serious brain damage
* ECT less than 3 months prior to this trial

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06; Primary Completion 2017-12 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Positive and Negative Symptom Scale | 2 days
  Positive and Negative Symptom Scale (PANSS) is assessed two days after ECT course

CONTACTS AND LOCATIONS:
Locations (1):
- Niuvanniemi Hospital, Kuopio, Finland